CLINICAL TRIAL: NCT06694766
Title: Comparative Study of Tolerance and Immunogenicity Induced by Primary Yellow Fever Vaccination in Pregnant and Non-pregnant Women
Brief Title: VAC-SIP-YF (Vaccination- Safety & Immunogenicity During Pregnancy- Yellow Fever)
Acronym: VAC-SIP-YF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Cerballiance (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-071; 2023-A02595-40 (Other: ID-RCB number)
Record Dates: First submitted 2024-10-14; First posted 2024-11-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Yellow Fever Vaccine
Keywords: Yellow Fever Vaccination Tolerance Immunogenicity Pregnancy

STUDY DESIGN:
Intervention Model Description: * women vaccinated during pregnancy
  * women vaccinated outside pregnancy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women vaccinated during pregnancy (Other): Participants who received a yellow fever vaccination during pregnancy
  Interventions: Procedure: Blood sample collection
- women vaccinated outside pregnancy (Other): Participants who received a yellow fever vaccination outside pregnancy
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — A blood sample collection of 18.5 mL will be required for the immunogenicity component.

SUMMARY:
The aim of this study is to compare the immunogenicity induced by yellow fever vaccination administered during pregnancy with that induced by vaccination outside pregnancy, and to assess the maternal and fetal tolerance of this vaccination.

DETAILED DESCRIPTION:
Yellow fever (YF), caused by the yellow fever virus (YFV), is an endemic disease in tropical and subtropical regions of South America and Africa. The virus is transmitted to humans by mosquitoes and can cause severe acute illness, leading to death in 20 to 60% of cases. There is currently no antiviral treatment available.

The yellow fever vaccine is a live attenuated virus vaccine recommended for individuals living in or traveling to tropical regions of Africa and South America. Under the International Health Regulations (IHR), cross-border travelers aged one year and older must present an immunization certificate issued by a government-approved international vaccination center. Globally, between twenty and sixty million doses are administered each year.

In France, the vaccine used against Yellow Fever is Stamaril® (Sanofi Pasteur MSD), which utilizes the 17D-204 strain. Due to insufficient data on the tolerance and immunogenicity induced by yellow fever vaccination during pregnancy, specific precautions and guidelines are recommended in this scenario. Currently, pregnancy is a relative contraindication for yellow fever vaccination. It may be considered for pregnant women who cannot postpone travel, are traveling to a yellow fever endemic area, and where the benefit-risk ratio of vaccination is deemed favorable by the attending physician.

This research consists of 2 sections:

* Tolerance section: related to yellow fever vaccination, will involve solely collecting retrospective data. This first component will be conducted during a telephone call led by the investigating physician.
* Immunogenicity section: to evaluate the immune response induced by yellow fever vaccination. This second component will be conducted during a visit to the CMIP, where a blood sample will be taken.

All women will participate in the tolerance assessment component. If they wish and sign the written consent, they may also participate in the immunogenicity assessment component. Following the telephone call, an appointment at the CMIP will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

Common :

* Person over 18 years of age at the time of the first yellow fever vaccination
* Female gender
* Oral consent obtained after subject has been informed
* Subject covered by Social Security with the exception of Aide Médicale d'Etat

Specific to both groups :

* For women vaccinated during pregnancy (case): Primary yellow fever vaccination during pregnancy
* For women vaccinated outside pregnancy (control): Primary yellow fever vaccination outside pregnancy

Exclusion Criteria:

Criteria common to both sections (tolerance and immunogenicity):

* Subject having received a second yellow fever vaccination
* Persons unable to give informed consent for participation
* Women born in areas where yellow fever is endemic
* Female adults under legal protection (guardianship or trusteeship)

Specific criteria for participants in the immunogenicity section:

* Medical condition imcompatible with 18.5 mL blood
* Women who have not given written consent to participate in the study. immunogenicity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 270 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Describe the immunogenicity induced by primary yellow fever vaccination during pregnancy and compare it to the immunogenicity induced by primary vaccination outside pregnancy | 36 months
  Proportion of participants with a neutralizing antibody rate above 1/10. A serological analysis will be performed to measure neutralizing antibody response by using PRNT 80 seroneutralization techniques.
  Each woman vaccinated against YF during pregnancy will be matched with a woman vaccinated outside pregnancy based on age (+/- 5 years) and time since primary YF vaccination (+/- 6 months).
  We anticipate that vaccination against YF during pregnancy will be equivalent in term of immunogenicity compared to vaccination against YF realized among non-pregnant women of the same age range. Based on the hypothesis of a protective immune response rate of 90% in the pregnant women group, a sample size in each group of 135, with a normal approximation test of proportions, will allow a type 1 risk of 0.05, a power of 80% and a minimum difference of 5%, in order to reject the null hypothesis according to which the protective immune response rates in the two groups are not equivalent.

SECONDARY OUTCOMES:
Describe the safety of yellow fever vaccination during pregnancy in women who have been vaccinated | 36 months
  The data collected for safety assessment regarding women will include:
  * Occurrence of YEL-AND or YEL-AVD
  * Local adverse effects (pain, oedema, erythema, satellite lymph node)
  * Nausea, vomiting, diarrhea, fever, arthralgia, myalgia
  * Other adverse events that occurred after vaccination
  All adverse reactions will be collected following MedDRA guidelines. The proportion of averse events will be compared to that of the non pregnant women group and to that of histoical series.
Describe the tolerability of yellow fever vaccination during pregnancy in the fetus and newborn. | 36 months
  Data collected for safety assessment regarding the fœtus and newborn will include :
  * Proportion of miscarriage, stillbirth, premature birth, and low weight birth and compare it to that of general population
  * From the infant health record:
  * Apgar, weight, size, and cranial perimeter at birth
  * Birth defect
  * Physical examination at birth (day 8), 9 month and 24 months of life
Create a biological collection for future studies on infectious/tropical diseases and the immune response to vaccination | 36 months
  This collection could allow :
  * analysis of cellular response to yellow fever vaccine e.g., activation of dendritic cells, NK cells, B lymphocytes and various T lymphocytes
  * exploration of participants' cellular immunity and identification of factors influencing the latter
  * Create a cohort of vaccinated women to assess immunogenicity and safety of all vaccines received during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Kaoutar JIDAR, MD, Principal Investigator — Medical Center of l'Institut Pasteur (CMIP)
Locations (1):
- Medical Center of Institut Pasteur, Paris, France